CLINICAL TRIAL: NCT07315919
Title: Integrating Planetary Health and Environmental Justice Into High School Construction Career Education: A Randomized Controlled Trial of the Ecosystem Justice Translator
Brief Title: Planetary Health and Environmental Justice in Construction Career Education
Acronym: EJT-CTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Devan Cantrell Addison-Turner, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-84369; DGE-2146755 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2025-12-20; First posted 2026-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Health Knowledge; Environmental Exposure; Attitude; Practice
Keywords: Environmental justice; Planetary health; Construction education; Workforce development; Health equity
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-Centered Design Curriculum with EJT (Experimental): 6-month Community-Centered Design curriculum integrating the Ecosystem Justice Translator (EJT). Structure: Weeks 1-4 foundations of planetary health and environmental justice; Weeks 5-10 EJT module training; Weeks 11-18 community engagement project with local stakeholder interviews; Weeks 19-24 capstone design project. Delivered during regular CTE class periods (~4 hours weekly). Students work in teams of 3-4 on authentic community challenges. EJT is a web-based computational system with four modules: Community Voice Equity Translation (CVET), Ecosystem Service Health Integration (ESHI), Environmental Justice Investment Prioritization (EJIP), and Uncertainty, Bias, and Risk Quantification (UBR).
  Interventions: Behavioral: Community-Centered Design Curriculum with EJT
- CONTROL (Active Comparator): Standard construction career curriculum per California CTE Model Curriculum Standards: building codes and permitting, construction safety (OSHA 10), blueprint reading and computer-aided design (CAD), materials science and selection, basic carpentry and framing. Control participants receive equal contact hours (~4 hours weekly for 24 weeks) without explicit health equity, environmental justice, or planetary health content. Control participants will be offered access to intervention materials and EJT software after study completion (waitlist control design).
  Interventions: Behavioral: Traditional Technical Curriculum

INTERVENTIONS:
Behavioral: Community-Centered Design Curriculum with EJT — 6-month (24-week) Community-Centered Design curriculum integrating the Ecosystem Justice Translator (EJT), delivered during regular CTE class periods (~4 hours weekly). EJT is a web-based computational system with four modules: (1) Community Voice Equity Translation using large language models; (2) Ecosystem Service Health Integration linking InVEST models with epidemiological dose-response functions; (3) Environmental Justice Investment Prioritization; (4) Uncertainty, Bias, and Risk Quantification. Curriculum structure: Weeks 1-4 planetary health foundations; Weeks 5-10 EJT training; Weeks 11-18 community engagement projects; Weeks 19-24 capstone design. Students work in teams of 3-4 on authentic community challenges.
  Other Names: Community-Centered Design Curriculum with Ecosystem Justice Translator; EJT Curriculum
  Arms: Community-Centered Design Curriculum with EJT
Behavioral: Traditional Technical Curriculum — Standard construction career curriculum per California CTE Model Curriculum Standards delivered over 24 weeks (~4 hours weekly). Content includes: building codes and permitting, construction safety (OSHA 10 certification), blueprint reading and CAD, materials science and selection, basic carpentry and framing techniques. Equal contact hours to intervention arm without explicit health equity, environmental justice, or planetary health content. Control participants offered access to EJT curriculum materials after study completion (waitlist control design).
  Arms: CONTROL

SUMMARY:
This study tests whether a new educational curriculum can help high school students in construction career programs better understand how building design affects community health and environmental justice. The study compares two approaches: (1) a new "Community-Centered Design" curriculum that uses the Ecosystem Justice Translator (EJT) software tool, which helps students see connections between construction decisions, energy efficiency, nature exposure, and health outcomes in different neighborhoods; versus (2) the traditional construction career curriculum that focuses on technical skills. Students aged 14-18 enrolled in construction career programs will be randomly assigned to one of these two groups. Over 6 months, the intervention group will learn to use the EJT tool and apply environmental justice concepts to construction projects. Researchers will measure how well students understand connections between construction, environment, and health at the start, middle, and end of the program, and again 6 months later. The goal is to determine if integrating environmental justice and health concepts into construction education improves students' awareness of how their future work can help or harm community health, particularly in disadvantaged neighborhoods.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18 years at enrollment
* Current enrollment in a participating construction career pathway program (minimum 2nd semester)
* Ability to participate in 6-month curriculum during regular CTE class periods
* Written informed consent from parent/guardian for participants under 18 years
* Written assent from student participant
* Ability to complete assessments in English (with accommodations as needed)

Exclusion Criteria:

* Prior participation in a formal environmental justice or planetary health curriculum within the past 12 months
* Expected inability to complete study assessments due to planned relocation or program withdrawal
* Concurrent enrollment in another research study involving educational interventions

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-08-05 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Health-Integrated Equity Consciousness Index (HI-ECI) | Baseline, 3 months, 6 months (primary endpoint), 12 months
  Composite measure of awareness of relationships between built environment, energy systems, nature exposure, and health equity. Derived from coded qualitative responses to standardized scenario prompts. Higher scores indicate greater health equity consciousness. Range 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Devan C. Addison-Turner, PhD in CEE, Principal Investigator — daddisonturner@stanford.edu
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
I may keep anonymous, unique Individual Participant Data (IPD) for participant performance tracking in a codebook and database. The information may be used to publish a journal paper.